CLINICAL TRIAL: NCT03538626
Title: VRC 609: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB091-00-AB (N6LS), Administered Intravenously or Subcutaneously With or Without Recombinant Human Hyaluronidase PH20 (rHuPH20) to Healthy Adults
Brief Title: Phase I, Open-Label, Dose-Escalation Study of a Human Monoclonal Antibody, VRC-HIVMAB091-00-AB (N6LS), Administered Intravenously or Subcutaneously With or Without Recombinant Human Hyaluronidase PH20 (rHuPH20)
Acronym: VRC 609
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180105; 18-I-0105
Record Dates: First submitted 2018-05-24; First posted 2018-05-29 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-12

CONDITIONS: HIV Antibodies
Keywords: Immune Cells; bNAb; Plasma Cell; HIV; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1: N6LS (5 mg/kg IV) single dose (Experimental): N6LS (5 mg/kg) administered by intravenous (IV) infusion (Day 0)
  Interventions: Biological: VRC-HIVMAB091-00-AB
- Group 2: N6LS (5 mg/kg SC) single dose (Experimental): N6LS (5 mg/kg) administered by subcutaneous (SC) injection (Day 0)
  Interventions: Biological: VRC-HIVMAB091-00-AB
- Group 3: N6LS (20 mg/kg IV) single dose (Experimental): N6LS (20 mg/kg) administered by IV infusion (Day 0)
  Interventions: Biological: VRC-HIVMAB091-00-AB
- Group 4: N6LS (40 mg/kg IV) single dose (Experimental): N6LS (40 mg/kg) administered by IV infusion (Day 0)
  Interventions: Biological: VRC-HIVMAB091-00-AB
- Group 5: N6LS (5 mg/kg SC) repeat dose (Experimental): N6LS (5 mg/kg) administered by SC injection (Day 0, Week 12 and Week 24)
  Interventions: Biological: VRC-HIVMAB091-00-AB
- Group 6: N6LS (20 mg/kg IV) repeat dose (Experimental): N6LS (20 mg/kg) administered by IV infusion (Day 0, Week 12 and Week 24)
  Interventions: Biological: VRC-HIVMAB091-00-AB
- Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) single dose (Experimental): N6LS (5 mg/kg) + rHuPH20 (2000 U/ml) administered by SC injection (Day 0)
  Interventions: Biological: VRC-HIVMAB091-00-AB; Biological: rHuPH20
- Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) single dose (Experimental): N6LS (20 mg/kg) + rHuPH20 (2000 U/ml) administered by SC injection (Day 0)
  Interventions: Biological: VRC-HIVMAB091-00-AB; Biological: rHuPH20

INTERVENTIONS:
Biological: VRC-HIVMAB091-00-AB — N6LS (VRC-HIVMAB091-00-AB) is a human monoclonal antibody targeted to the HIV-1 CD4 binding site.
Biological: rHuPH20 — Recombinant human hyaluronidase PH20 (rHuPH20) is the active ingredient of the investigational ENHANZE™ Drug Product (EDP). EDP is a purified preparation of rHuPH20.
  Other Names: EDP
  Arms: Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) single dose; Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) single dose

SUMMARY:
Background:

The experimental product in this study, N6LS, is a human monoclonal antibody. Antibodies are one way that the human body fights infection. Monoclonal means that all the antibodies in the product are the same. N6LS is directed against the HIV virus. There is no HIV in the N6LS study product and you cannot get HIV from this product. This study is the first time N6LS is tested in humans. It was given into a vein in the arm (intravenously, IV) or as an injection underneath the skin (subcutaneously, SC). The study also tested N6LS mixed with an enzyme, rHuPH20 (recombinant human hyaluronidase). rHuPH20 increases the spread of fluids injected underneath your skin (subcutaneously, SC) and allows for the rapid delivery of large volume injections that can be given with a single needle. It was given as a SC infusion using a small needle attached to an infusion pump. Study products were only given to healthy adults who are not infected with HIV.

Objective:

The main purpose of the study is to see if N6LS alone and N6LS mixed with rHuPH20 is safe in healthy adults. Another goal is to learn how amounts of N6LS in the body change over time.

Study Plan:

Assigned study groups depended on the dose of product, the numbers of times the product was given (once or three times at 12-week intervals), and how the product was given (IV or SC). Blood samples for research were collected at most of the visits. There were about 14 clinic visits over 6 months for all groups who got one dose of product, and about 26 clinic visits over 12 months for the groups who got three doses of product.

DETAILED DESCRIPTION:
Study Design:

This is the first study in healthy adults of the N6LS monoclonal antibody (MAb). It was a dose-escalation study to examine safety, tolerability, dose, and pharmacokinetics (PK) of N6LS administered intravenously (IV) and subcutaneously (SC) to healthy adults. For SC administration, N6LS was administered alone or co-administered with the permeation enhancer rHuPH20 enzyme. Primary hypotheses are that N6LS administration to healthy adults will be safe by the IV and SC routes, alone and with rHuPH20 co-administration. A secondary hypothesis is that all N6LS administrations will be detectable in human sera with a definable half-life

Product Description:

N6LS (VRC-HIVMAB091-00-AB) is a human MAb targeted to the HIV-1 CD4 binding site. It was developed by the VRC/NIAID/NIH and manufactured under current Good Manufacturing Practice (cGMP) regulations at the VRC Vaccine Pilot Plant operated under contract by the Vaccine Clinical Materials Program (VCMP), Leidos Biomedical Research, Inc., Frederick, MD. The product was provided as a sterile aqueous buffered solution in 10 mL glass vials at a concentration of 100 mg/mL and volume of 6.25 mL.

Each vial of ENHANZE™ Drug Product (EDP) contains 0.5 mL of rHuPH20 formulated at a concentration of 1 mg/mL (approximately 110,000 U/mL rHuPH20). rHuPH20 is a tissue permeability modifier that depolymerizes hyaluronan (HA), increasing the dispersion of a substance into the subcutaneous space, which enables SC delivery of co-administered antibody (-ies) at higher dose volumes (e.g., >10 mL) that cannot be administered quickly without rHuPH20. EDP is manufactured by Ajinomoto Althea, Inc. (San Diego, CA) for Halozyme Therapeutics, Inc. (San Diego, CA) and is supplied in 2 mL glass vials as a sterile, single-dose, injectable liquid.

Subjects:

Healthy adults, 18-50 years of age.

Study Plan:

This open-label study included 8 dose groups to assess N6LS alone given as a single IV infusion at the 5, 20, or 40 mg/kg dose level (Groups 1,3 and 4); a single SC injection at the 5 mg/kg dose level (Group 2); or in 3 administrations, spaced 12 weeks apart by SC injection at the 5 mg/kg dose level (Group 5), or by IV infusion at the 20 mg/kg dose level (Group 6). Two additional groups assessed N6LS given as a single SC injection mixed with rHuPH20 (2000 U/mL) at 5 mg/kg (Group 7) or 20 mg/kg (Group 8) doses. Enrollment opened with Groups 1, 2 and 5; and was followed by the sequential activation of Groups 3, 4, and 6. With implementation of the two SC N6LS+rHuPH20 arms as a protocol amendment, Group 7 opened first to accrual, followed by Group 8.

Study Duration:

Study participation was approximately 24 weeks for participants in Groups 1-4, 7 and 8; and 48 weeks for participants in Groups 5 and 6.

ELIGIBILITY:
INCLUSION CRITERIA:

A volunteer must have met all of the following criteria:

1. Willing and able to complete the informed consent process.
2. 18 to 50 years of age.
3. Based on history and examination, must be in good general health and without history of any of the conditions listed in the exclusion criteria.
4. Willing to have blood samples collected, stored indefinitely, and used for research purposes.
5. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
6. Screening laboratory criteria within 84 days prior to enrollment meeting the following criteria:

   * White blood cell count (WBC): 2,500-12,000/mm^3.
   * WBC differential: Within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
   * Platelets: 125,000-400,000/mm^3.
   * Hemoglobin: Within institutional normal range or accompanied by PI or designee approval.
   * Creatinine: less than or equal to 1.1 x Upper Limit of Normal (ULN).
   * Alanine aminotransferase (ALT): less than or equal to 1.25 x ULN.
   * Aspartate aminotransferase (AST): less than or equal to 1.25 x ULN.
   * Negative for HIV infection by an FDA approved method of detection.

   Female-Specific Criteria:
7. If a woman is of reproductive potential and sexually active with a male partner, then she agrees to use an effective means of birth control from the time of study enrollment until the last study visit, or to be monogamous with a partner who has had a vasectomy.
8. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A volunteer would have been excluded if one or more of the following conditions applied:

1. Prior receipt of licensed or investigational monoclonal antibody.
2. Weight > 115 kg.
3. Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis within the 2 years prior to enrollment that has a reasonable risk of recurrence during the study.
4. Hypertension that is not well controlled.
5. Woman who is breast-feeding, or planning to become pregnant during the study participation.
6. Receipt of any investigational study agent within 28 days prior to enrollment.
7. Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the subject including (but not limited to): diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of drug or alcohol abuse, asthma, autoimmune disease, infectious disease, psychiatric disorders, heart disease, or cancer.
8. Known hypersensitivity to hyaluronidase or any of the excipients in ENHANZE™ Drug Product (EDP).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wu, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not shared because it has limited value in a small phase 1 trial of healthy volunteers. We instead report non-IPD data as required in ClinicalTrials.gov.

REFERENCES:
- [Background] Huang J, Kang BH, Ishida E, Zhou T, Griesman T, Sheng Z, Wu F, Doria-Rose NA, Zhang B, McKee K, O'Dell S, Chuang GY, Druz A, Georgiev IS, Schramm CA, Zheng A, Joyce MG, Asokan M, Ransier A, Darko S, Migueles SA, Bailer RT, Louder MK, Alam SM, Parks R, Kelsoe G, Von Holle T, Haynes BF, Douek DC, Hirsch V, Seaman MS, Shapiro L, Mascola JR, Kwong PD, Connors M. Identification of a CD4-Binding-Site Antibody to HIV that Evolved Near-Pan Neutralization Breadth. Immunity. 2016 Nov 15;45(5):1108-1121. doi: 10.1016/j.immuni.2016.10.027. PMID 27851912
- [Background] Gaudinski MR, Coates EE, Houser KV, Chen GL, Yamshchikov G, Saunders JG, Holman LA, Gordon I, Plummer S, Hendel CS, Conan-Cibotti M, Lorenzo MG, Sitar S, Carlton K, Laurencot C, Bailer RT, Narpala S, McDermott AB, Namboodiri AM, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Graham BS, Mascola JR, Ledgerwood JE; VRC 606 Study Team. Safety and pharmacokinetics of the Fc-modified HIV-1 human monoclonal antibody VRC01LS: A Phase 1 open-label clinical trial in healthy adults. PLoS Med. 2018 Jan 24;15(1):e1002493. doi: 10.1371/journal.pmed.1002493. eCollection 2018 Jan. PMID 29364886
- [Background] Ledgerwood JE, Coates EE, Yamshchikov G, Saunders JG, Holman L, Enama ME, DeZure A, Lynch RM, Gordon I, Plummer S, Hendel CS, Pegu A, Conan-Cibotti M, Sitar S, Bailer RT, Narpala S, McDermott A, Louder M, O'Dell S, Mohan S, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Mascola JR, Graham BS; VRC 602 Study Team. Safety, pharmacokinetics and neutralization of the broadly neutralizing HIV-1 human monoclonal antibody VRC01 in healthy adults. Clin Exp Immunol. 2015 Dec;182(3):289-301. doi: 10.1111/cei.12692. Epub 2015 Sep 24. PMID 26332605
- [Derived] Wu RL, Houser KV, Gaudinski MR, Widge AT, Awan SF, Carter CA, Holman LA, Saunders J, Hendel CS, Eshun A, Whalen WR, Wang X, Arthur A, Cunningham JE, Beck A, Casazza JP, Yamshchikov GV, Rothwell RS, Strom L, Dittakavi T, Happe M, Hickman SP, Conan-Cibotti M, Carlton K, Zhang L, Huang Y, Capparelli EV, Castro M, Lin BC, O'Connell S, Flach BS, Bailer RT, Narpala SR, Serebryannyy L, McDermott AB, Arnold FJ, Gall JG, Vazquez S, Berkowitz NM, Gordon IJ, Chen GL, Kwong PD, Huang J, Pierson TC, Connors M, Mascola JR, Zhou T, Doria-Rose NA, Koup RA, Dropulic LK; VRC 609 study team. Safety and pharmacokinetics of N6LS, a broadly neutralising monoclonal antibody for HIV: a phase 1, open-label, dose-escalation study in healthy adults. Lancet HIV. 2025 Jul;12(7):e485-e495. doi: 10.1016/S2352-3018(25)00041-4. Epub 2025 May 20. PMID 40409326
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-I-0105.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited for the study at the NIH Clinical Center in Bethesda, Maryland, USA.
Period: Overall Study
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Started | 3 | 4 | 3 | 3 | 5 | 5 | 5 | 5
Received First Product Administration | 3 | 3 (One Group 2 participant withdrew from the study prior to product administration.) | 3 | 3 | 5 | 5 | 5 | 5
Received All Product Administrations | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Completed | 3 | 3 | 3 | 3 | 5 | 5 | 4 (One Group 7 participant was lost to follow up after the product administration was completed.) | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population included all enrolled participants. Weight represents weight at time of enrollment. Age represents age at enrollment day.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 5 | 5 | 5 | 5 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] — Age represents age at enrollment day.
  years | 30.3 (7.4) | 31.3 (7.4) | 29.0 (6.6) | 28.0 (7.8) | 31.0 (8.5) | 26.2 (7.8) | 37.6 (12.5) | 32.8 (12.0) | 31.1 (9.0)
Age, Customized [Count of Participants; unit: Participants] — Age represents age at enrollment day.
  Participants
    21-30 years | 1 | 2 | 2 | 2 | 2 | 4 | 2 | 3 | 18
    31-40 years | 2 | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 10
    41-50 years | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 2 | 4 | 3 | 2 | 3 | 19
  Male | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 3 | 4 | 2 | 2 | 5 | 5 | 4 | 5 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 4
  White | 1 | 2 | 3 | 2 | 2 | 3 | 3 | 4 | 20
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Weight (kg) [Mean (Standard Deviation); unit: kg] — Weight represents weight at time of enrollment.
  kg | 79.9 (16.0) | 88.5 (17.1) | 90.7 (3.2) | 61.7 (11.8) | 82.0 (15.3) | 74.7 (13.8) | 83.9 (5.6) | 73.4 (9.3) | 79.4 (13.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 3 Days of N6LS Product Administration Alone or N6LS Co-Administered With rHuPH20
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 3 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 3 days after each product administration, at approximately Day 3 for all dose groups, and at approximately Day 87 and Day 171 for repeat dose groups
Population: Population included all enrolled participants who received at least one dose of study product and provided safety data (via diary card). One participant in Group 2 withdrew from the study prior to receiving study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Participants
  Pain/Tenderness: None | 3 | 1 | 3 | 3 | 1 | 5 | 3 | 1
  Pain/Tenderness: Mild | 0 | 2 | 0 | 0 | 4 | 0 | 2 | 3
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: None | 3 | 3 | 3 | 3 | 5 | 4 | 5 | 5
  Bruising: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: Moderate | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 4
  Swelling: Mild | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 3 | 3 | 3 | 3 | 3 | 5 | 0 | 0
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1
  Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
  Pruritis (Itching): None | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 2
  Pruritis (Itching): Mild | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
  Pruritis (Itching): Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Pruritis (Itching): Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 3 | 1 | 3 | 3 | 1 | 4 | 0 | 0
  Any Local Symptom: Mild | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 3 Days of N6LS Product Administration Alone or N6LS Co-Administered With rHuPH20
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 3 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Participants
  Malaise: None | 3 | 3 | 2 | 3 | 4 | 5 | 5 | 4
  Malaise: Mild | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Malaise: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 3 | 3 | 3 | 3 | 4 | 5 | 5 | 5
  Myalgia: Mild | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 2 | 3 | 1 | 2 | 4 | 5 | 5 | 5
  Headache: Mild | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
  Headache: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 3 | 3 | 3 | 2 | 5 | 5 | 5 | 5
  Chills: Mild | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 3 | 3 | 3 | 2 | 4 | 5 | 5 | 4
  Nausea: Mild | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): None | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
  Temperature (Fever): Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
  Joint Pain: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 2 | 3 | 1 | 2 | 2 | 5 | 5 | 3
  Any Systemic Symptom: Mild | 1 | 0 | 2 | 1 | 3 | 0 | 0 | 2
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following N6LS Product Administration Alone or N6LS Co-Administered With rHuPH20
Description: Unsolicited adverse event (AE) data collection included AEs of all severities from the date of product administration through the Day 56 (8 weeks) after each product administration visit. After the Day 56 (8 weeks) after each product administration visit, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions that require ongoing medical management (reported as a separate outcome) were recorded through the last study visit. The relationship between a non-serious AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 8 weeks after each product administration, at approximately Week 8 for all dose groups, and at Weeks 20 and 32 for repeat dose groups
Population: Population included all enrolled participants who received at least one dose of study product and had safety data collected (via clinical assessment and/or lab results). One participant in Group 2 withdrew from the study prior to receiving study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Participants
  Related to Study Product | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 1
  Unrelated to Study Product | 1 | 1 | 1 | 2 | 2 | 3 | 2 | 2
  Total Number of Participants who had One or More Non-Serious Unsolicited AE | 1 | 3 | 2 | 2 | 3 | 5 | 2 | 3

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following N6LS Product Administration Alone or N6LS Co-Administered With rHuPH20
Description: SAEs were recorded from receipt of first study product administration through the last expected study visit at Week 24 for single dose groups and at Week 48 for repeat dose groups. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after product administration through the study participation, up to Week 24 for single dose groups and up to Week 48 for repeat dose groups
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following N6LS Product Administration Alone or N6LS Co-Administered With rHuPH20
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of first study product administration through the last expected study visit at Week 24 for single dose groups and at Week 48 for repeat dose groups. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following N6LS Product Administration Alone or N6LS Co-Administered With rHuPH20
Description: Abnormal laboratory results recorded as unsolicited adverse events (AEs) are summarized. Safety lab parameters included hematology (hemoglobin, hematocrit, mean corpuscular volume (MCV) platelets, and neutrophil, lymphocyte, monocyte, eosinophil and basophil counts) and chemistry (alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine, alkaline phosphatase (ALP) and Comprehensive Metabolic Panel (CMP)). Complete Blood Count (CBC) with differential and chemistry (ALT, AST, ALP, creatinine and CMP) results were collected at different timepoints throughout the study per the protocol's schedule of evaluations. Institutional laboratory normal ranges as well as the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 were used.
Time Frame: as for outcome 3
Population: Population included all enrolled participants who received at least one dose of study product and had safety data collected via laboratory results. One participant in Group 2 withdrew from the study prior to receiving study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Participants
  Neutrophil Count | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase (ALT) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Aspartate aminotransferase (AST) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Creatinine | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Number of Participants with one or more Abnormal Laboratory Results AE Related to Study Product | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Number of Participants with one or more Abnormal Laboratory Results AE Unrelated to Study Product | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 0

7. Secondary Outcome: Number of Participants Who Produced N6LS Anti-drug Antibodies (ADA) Following N6LS Product Administration Alone or N6LS Co-Administered With rHuPH20
Description: A three-tiered assay was used for ADA evaluation. The tier 1 screening assay measures specific and non-specific binding of serum proteins to N6LS. The tier 2 assay is a qualitative competition assay in which exogenously added N6LS removes any N6LS-binding proteins from the serum prior to the binding assay. If the addition of the exogenous N6LS results in a reduction of signal, the specificity of N6LS binding is confirmed. The tier 3 assay is a qualitative assay that assesses the ability of N6LS-binding serum protein to prevent N6LS-mediated neutralization of an HIV pseudovirus in vitro. Only samples positive for a tier were analyzed in subsequent tiers.
Time Frame: Baseline and Weeks 4 and 8 for single dose groups, or Baseline and Weeks 4, 28, and 32 for repeat dose groups
Population: Population included all enrolled participants who received at least one dose of study product with up to 8 weeks of pharmacokinetic data for single dose groups (1-4 and 7-8, N=22) and up to 32 weeks of pharmacokinetic data for repeat dose groups (5-6, N=10). One participant in Group 2 withdrew from the study prior to receiving study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Participants
  Tier 1 ADA-Positive Sample | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 0
  Tier 2 ADA-Positive Sample | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Tier 3 ADA-Positive Sample | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

8. Secondary Outcome: Pharmacokinetic (PK) Parameters of N6LS: Maximum Observed Serum Concentration (Cmax)
Description: Cmax is the peak serum concentration that N6LS achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group.
Time Frame: Baseline through the study participation, up to Week 24 for single dose groups and up to Week 48 for repeat dose groups
Population: Population included all enrolled participants who received at least one dose of study product with up to 24 weeks of pharmacokinetic data for single dose groups (1-4 and 7-8, N=22) and up to 48 weeks of pharmacokinetic data for repeat dose groups (5-6, N=10). One participant in Group 2 withdrew from the study prior to receiving study product.
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
μg/ml | 109.0 (28.6) | 20.8 (1.9) | 492.7 (22.9) | 737.3 (53.7) | 21.3 (5.4) | 411.0 (76.7) | 37.3 (3.9) | 108.8 (40.6)

9. Secondary Outcome: Pharmacokinetic (PK) Parameters of N6LS: Time to Reach Maximum Observed Serum Concentration (Tmax)
Description: Tmax is the time it takes to reach Cmax of N6LS after it has been administered; it is determined based on the summary PK curve for each dose group.
Time Frame: Baseline through the study participation, up to Week 24 for single dose groups and up to Week 48 for repeat dose groups
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
days | 0.12 (0.05) | 2.85 (1.02) | 0.12 (0.09) | 0.13 (0.07) | 6.87 (0.07) | 0.03 (0.02) | 2.56 (0.44) | 4.34 (2.38)

10. Secondary Outcome: Pharmacokinetic (PK) Parameters of N6LS: Beta Half-life (T1/2b)
Description: Beta half-life (T1/2b) will be reported for this study. Beta half-life (T1/2b) is the time required for half of the N6LS product to be eliminated from the serum.
Time Frame: Baseline through the study participation, up to Week 24 for single dose groups and up to Week 48 for repeat dose groups
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
days | 48.7 (3.5) | 46.8 (1.7) | 50.9 (2.3) | 45.3 (4.4) | 49.9 (4.6) | 46.9 (1.9) | 49.2 (2.0) | 49.8 (6.5)

11. Secondary Outcome: Pharmacokinetic (PK) Parameters of N6LS: Clearance Rate
Description: Clearance is the rate of N6LS elimination divided by the plasma N6LS concentration; determined based on the summary pharmacokinetic (PK) curve for each study group. Clearance following a SC administration is calculated as Clearance (CL)/Bioavailability (F).
Time Frame: Baseline through the study participation, up to Week 24 for single dose groups and up to Week 48 for repeat dose groups
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ml/day
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
ml/day | 143.1 (35.1) | 365.3 (108.5) | 142.3 (13.3) | 131.0 (22.7) | 297.6 (60.3) | 148.3 (28.3) | 205.9 (16.8) | 253.7 (102.0)

12. Secondary Outcome: Pharmacokinetic (PK) Parameters of N6LS: Volume of Distribution
Description: Theoretical volume that would be necessary to contain the total amount of administered drug at the same concentration as observed in plasma. It represents the degree to which a drug is distributed in body tissue rather than the plasma and calculated based in the PK curve for each study group. Volume of distribution following a SC administration is calculated as Volume of distribution (V)/Bioavailability (F).
Time Frame: Baseline through the study participation, up to Week 24 for single dose groups and up to Week 48 for repeat dose groups
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5
Liter | 9.6 (2.6) | 23.2 (6.5) | 9.9 (0.4) | 7.9 (1.2) | 20.5 (2.6) | 9.3 (1.5) | 13.5 (0.9) | 16.6 (5.6)

ADVERSE EVENTS:
Time Frame: Unsolicited adverse event (AE) data collection included AEs of all severities after each study product administration through the Day 56 (8 weeks) visit. After the Day 56 visit, only serious AEs (SAEs) and new chronic medical conditions that required ongoing medical management were recorded through the study participation, up to Week 24 for single dose groups (1-4 and 7-8, N=22) and up to Week 48 for repeat dose groups (5-6, N=10).
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: N6LS (5 mg/kg IV) Single Dose | Group 2: N6LS (5 mg/kg SC) Single Dose | Group 3: N6LS (20 mg/kg IV) Single Dose | Group 4: N6LS (40 mg/kg IV) Single Dose | Group 5: N6LS (5 mg/kg SC) Repeat Dose | Group 6: N6LS (20 mg/kg IV) Repeat Dose | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 3/3 | 2/3 | 5/5 | 5/5 | 5/5 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: N6LS (5 mg/kg IV) Single Dose (N=3) | Group 2: N6LS (5 mg/kg SC) Single Dose (N=3) | Group 3: N6LS (20 mg/kg IV) Single Dose (N=3) | Group 4: N6LS (40 mg/kg IV) Single Dose (N=3) | Group 5: N6LS (5 mg/kg SC) Repeat Dose (N=5) | Group 6: N6LS (20 mg/kg IV) Repeat Dose (N=5) | Group 7: N6LS (5 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose (N=5) | Group 8: N6LS (20 mg/kg SC) + rHuPH20 (2000 U/ml SC) Single Dose (N=5)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1
Administration site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Biopsy (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biopsy breast (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sebaceous cyst excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Administration site pain (General disorders) | 0 | 2 | 0 | 0 | 4 | 0 | 2 | 4
Administration site pruritus (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Administration site swelling (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Administration site erythema (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 5
Administration site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT03538626/Prot_SAP_ICF_000.pdf